CLINICAL TRIAL: NCT03116672
Title: The Outcome of Preoperative Administration of Single-dose Ketorolac, Non-steroidal Anti-inflammatory Drug and Placebo on Postoperative Pain in Teeth With Irreversible Pulpitis and Apical Periodontitis
Brief Title: The Outcome of Preoperative Administration of Single-dose Ketorolac, Non-steroidal Anti-inflammatory Drug and Placebo
Acronym: PreOp
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Jorge Paredes Vieyra, Principal Investigator. PhD, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: One Dose 2017
Record Dates: First submitted 2017-03-28; First posted 2017-04-17 (Actual); Last update posted 2017-04-18 (Actual); Status verified 2017-04

CONDITIONS: Pulpitis - Irreversible
Keywords: pain; Diclofenac; NSAID; Ketorolac
MeSH Terms: conditions — Pain | interventions — Ketorolac; Diclofenac

STUDY DESIGN:
Intervention Model Description: Patient selection.
  Fifty-four of sixty-five patients (29 women and 25 men), 18 to 60 years of age with 54 eligible teeth consented to participate in the study. The patients were randomly divided into three groups using a web program. The patient number and group number were recorded. Informed consent was obtained from each patient and the possible discomforts and risks were fully explained.
  A total of 54 patients were divided into three groups (n = 18) according to the type of preoperative drug administrated.
Who Masked: Participant
Masking Description: Patient selection.
  Fifty-four of sixty-five patients (29 women and 25 men), 18 to 60 years of age with 54 eligible teeth consented to participate in the study. The patients were randomly divided into three groups using a web program. The patient number and group number were recorded. Informed consent was obtained from each patient and the possible discomforts and risks were fully explained.
  A total of 54 patients were divided into three groups (n = 18) according to the type of preoperative drug administrated, as follows: Group A: Administration of ketorolac 10mg, Group B: Administration of Diclofenac Na 50mg, and Group C: A placebo (capsule filled with sugar).
  After 15 minutes each participant received the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ketorolac 10 mg (Experimental): Administration of one dose Ketorolac 10 mg 15 minutes before treatment
  Interventions: Drug: one dose ketorolac 10 mg
- Diclofenac (Experimental): Administration of one dose Diclofenac 15 minutes before treatment
  Interventions: Drug: One dose Diclofenac
- Placebo oral capsule (Experimental): Administration of Placebo capsule 15 minutes before treatment
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: one dose ketorolac 10 mg — Administration of ketorolac 10mg, (Dolac) 15 minutes before the clinical procedure.
  Other Names: Dolac
  Arms: ketorolac 10 mg
Drug: One dose Diclofenac — Administration of diclofenac, (Diclofenaco) 15 minutes before the clinical procedure.
  Other Names: Diclofenaco
  Arms: Diclofenac
Drug: Placebo oral capsule — Administration of Placebo, 15 minutes before the clinical procedure.
  Other Names: Placebo OS
  Arms: Placebo oral capsule

SUMMARY:
Aim. To compare the outcome of preoperative administration of single-dose ketorolac, non-steroidal anti-inflammatory drug and placebo on postoperative pain in teeth with irreversible pulpitis and apical periodontitis.

DETAILED DESCRIPTION:
The institutional review board of the Faculty od Odontology Tijuana México approved the study protocol and all the participants were treated in accordance with the Helsinki Declaration (www.cirp.org/library/ethics/helsinki). The study started in February 2016 and ended in February 2017. The main inclusion criteria were: a) A diagnosis of pulpitis confirmed by positive response to hot and cold tests and b) Clinical and radiographic evidence of symptomatic apical periodontitis. It was determined based on the clinical symptoms severe preoperative pain (VAS > 60) and severe percussion pain (VAS > 60). Confirmed by positive response to hot and cold tests. Thermal pulp testing was performed by the author, and radiographic interpretation was verified by one certified oral surgeon.

Patient selection.

Fifty-four of sixty-five patients (29 women and 25 men), 18 to 60 years of age with 54 eligible teeth consented to participate in the study. The study design is shown in Figure 1. The patients were randomly divided into three groups using a web program. The patient number and group number were recorded. Informed consent was obtained from each patient and the possible discomforts and risks were fully explained.

A total of 54 patients were divided into three groups (n = 18) according to the type of preoperative drug administrated, as follows: Group A: ketorolac 10mg (Siegfried Rhein S.A. de C.V, Mexico,DF), Group B: Diclofenac Na 50mg (Voltaren, Novartis Mexico), and Group C: A placebo (capsule filled with sugar).

A registered pharmacist compounded identical-appearing capsules of the ketorolac, Diclofenac Na and the placebo (opaque yellow size ''0'' capsules). All medications were placed in identical bottles so that they were indistinguishable to the investigator.

The administration of drugs and root canal treatment were performed by two different researchers. One assistant knew the allocation and the drug type in the capsules, but the operator and the patient did not know which drug type was administered.

Patient selection was based on the following criteria: 1) The aims and requirements of the study were freely accepted; 2) Treatment was limited to patients in good health; 3) Patients with symptomatic or asymptomatic teeth with vital pulps and apical periodontitis; 4) A positive response to hot and cold pulp sensitivity tests; 5) Presence of sufficient coronal tooth structure for rubber dam isolation; 6) No prior endodontic treatment on the involved tooth and 7) No analgesics or antibiotics were used five days before the clinical procedures began.

Exclusion criteria included the following: 1) Patients who did not meet inclusion requirements; 2) Patients who did not provide authorization for participation; 3) Patients who were younger than 16 years old; 4) Patients who were pregnant; 5) Patients who were diabetic; 6) Patients with a positive history of antibiotic use within the past month; 7) Patients whose tooth had been previously accessed or endodontically treated; 8) Teeth with root resorption, and 9) Immature/open apex, or a root canal in which patency of the apical foramen could not be established were all excluded from the study. Teeth with periodontal pockets deeper than 4 mm, or the presence of a periapical radiolucency more than 2 cm diameter also were excluded of the study.

ELIGIBILITY:
Inclusion Criteria:

Patient selection was based on the following criteria:

1. The aims and requirements of the study were freely accepted;
2. Treatment was limited to patients in good health;
3. Patients with symptomatic or asymptomatic teeth with vital pulps and apical periodontitis;
4. A positive response to hot and cold pulp sensitivity tests;
5. Presence of sufficient coronal tooth structure for rubber dam isolation;
6. No prior endodontic treatment on the involved tooth and
7. No analgesics or antibiotics were used five days before the clinical procedures began.

Exclusion Criteria:

Exclusion criteria included the following:

1. Patients who did not meet inclusion requirements;
2. Patients who did not provide authorization for participation;
3. Patients who were younger than 16 years old;
4. Patients who were pregnant;
5. Patients who were diabetic;
6. Patients with a positive history of antibiotic use within the past month;
7. Patients whose tooth had been previously accessed or endodontically treated;
8. Teeth with root resorption, and
9. Immature/open apex, or a root canal in which patency of the apical foramen could not be established were all excluded from the study. Teeth with periodontal pockets deeper than 4 mm, or the presence of a periapical radiolucency more than 2 cm diameter also were excluded of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 3 (Actual)
Dates: Start 2016-02-02 (Actual); Primary Completion 2017-02-06 (Actual); Study Completion 2017-02-10 (Actual)

PRIMARY OUTCOMES:
Level of post operative pain with administration of single-dose ketorolac, non-steroidal anti-inflammatory drug and placebo on postoperative pain in teeth with irreversible pulpitis and apical periodontitis | 1 year after RCT
  One dose administration before the RCT done

SECONDARY OUTCOMES:
Level of Post operative pain after administration of single dose before RCT | One year after root canal treatment
  One dose of placebo

CONTACTS AND LOCATIONS:
Overall Officials: Miguel O Osuna, DDS, Study Director — SECRETARIA DE SALUD DE BC
Locations (1):
- Jose Clemente, Tijuana, Estado de Baja California, Mexico

IPD SHARING:
Plan to Share IPD: Yes
Invitation to participate. Offer to the public All the clinical procedure and risks were explained to each participant.

REFERENCES:
- [Result] Paredes-Vieyra J, Enriquez FJ. Success rate of single- versus two-visit root canal treatment of teeth with apical periodontitis: a randomized controlled trial. J Endod. 2012 Sep;38(9):1164-9. doi: 10.1016/j.joen.2012.05.021. Epub 2012 Jul 26. PMID 22892729
- Available data/document: Clinical Study Report: UABC — http://www.uabc.mx — Clinical trial that evaluate drug and placebo
- Available data/document: Individual Participant Data Set: protocol guide — http://www.uabc.mx — Clinical Guide